CLINICAL TRIAL: NCT06606990
Title: Pilot Study of Pidnarulex Pharmacodynamics in Patients With Advanced Solid Tumors
Brief Title: Testing How the Body Responds to the Drug CX-5461 (Pidnarulex) in Patients With Metastatic Solid Cancers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2024-07701; NCI-2024-07701 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); IRB002354; IRB002325; 10667 (Other: National Cancer Institute LAO); 10667 (Other: CTEP)
Record Dates: First submitted 2024-09-20; First posted 2024-09-23 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Malignant Solid Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Biopsy; Specimen Handling; Magnetic Resonance Spectroscopy; CX 5461

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (pidnarulex) (Experimental): Patients receive pidnarulex IV over 60 minutes on days 1 and 8 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT or MRI, biopsy, and collection of blood samples throughout the trial. Patients may undergo ECHO at screening and then as clinically indicated.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Echocardiography Test; Procedure: Magnetic Resonance Imaging; Biological: Pidnarulex

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Biological: Pidnarulex — Given IV
  Other Names: CX-5461; CX5461; Pol I Inhibitor CX5461; RNA Pol I Inhibitor CX5461

SUMMARY:
This phase I trial tests the safety, side effects, and best dose of pidnarulex (CX-5461) in treating patients with solid tumors that have spread from where it first started (primary site) to other places in the body (metastatic). Pidnarulex is an oral inhibitor of ribonucleic acid polymerase I, with potential antineoplastic activity. It blocks a certain enzyme needed for cell division and deoxyribonucleic acid (DNA) repair and may kill cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess whether pidnarulex induces a Rad51 response, which will be determined by an integral biomarker of percentage of cells with Rad51 nuclear foci in tumor biopsy specimens in patients with and without homologous repair deficiency (HRD) genetic mutations.

SECONDARY OBJECTIVES:

I. To determine the safety and tolerability of pidnarulex. II. To determine the overall response rate (complete responses plus partial responses) in patients with advanced, refractory solid tumors.

III. To measure the pharmacokinetics of pidnarulex. IV. To evaluate other DNA damage and repair signaling markers including Top2, G4 stabilization, RPA32, pSer33-RPA32, γH2AX, 53BP1, pSer8-RPA32, pKap1m and pNBS1.

EXPLORATORY OBJECTIVE:

I. To examine genomic alterations in circulating tumor DNA (ctDNA) that may be associated with response or resistance.

OUTLINE:

Patients receive pidnarulex intravenously (IV) over 60 minutes on days 1 and 8 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo computed tomography (CT) or magnetic resonance imaging (MRI), biopsy, and collection of blood samples throughout the trial. Patients may undergo echocardiography (ECHO) at screening and then as clinically indicated.

After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed solid tumors with metastatic disease that have progressed after ≥ 1 line of prior therapy and/or for whom no standard treatment is available that has been shown to improve survival.
* Patients must have a molecular testing report to assess HRD mutation status prior to enrollment.
* Patients must have measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1, with at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥ 20 mm (≥ 2 cm) by chest x-ray or as ≥ 10 mm (≥ 1 cm) with CT scan, MRI, or calipers by clinical exam).
* Patients must have a tumor site amenable to biopsy.
* Age ≥ 18 years of age.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2 (Karnofsky ≥ 70%).
* Absolute neutrophil count ≥ 1,500/mcL.
* Hemoglobin ≥ 9 g/dL.
* Platelets ≥ 100,000/mcL.
* Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN).

  * (However, patients with known Gilbert disease who have serum bilirubin level of up to 3 mg/dl may be enrolled).
* International normalized ratio (INR) or activated partial thromboplastin time (aPTT) ≤ 1.5 institutional upper limit of normal (ULN).

  * Subjects may receive supplementation to meet this eligibility criteria.
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic-pyruvic transaminase [SGPT]) ≤ 3 x institutional ULN.

  * (AST and/or ALT ≤ 5 x ULN for patients with liver involvement).
* Potassium ≥ lower limit of normal (LLN).

  * Subjects may receive supplementation to meet this eligibility criteria.
* Magnesium ≥ LLN.

  * Subjects may receive supplementation to meet this eligibility criteria.
* Ionized or corrected calcium ≥ LLN.

  * Subjects may receive supplementation to meet this eligibility criteria.
* Creatinine ≤ 1.5 x institutional ULN OR creatinine clearance levels ≥ 60 ml/min based on the Cockcroft-Gault formula.
* Oxygen (O2) saturation > 90% on room air.
* Prior standard or investigational therapy must have been completed ≥ 4 weeks or ≥ 5 half-lives of the prior agent (whichever is shorter) prior to enrollment; the exception is ≥ 2 weeks since any investigational agent administered (at a sub-therapeutic dose) as part of a phase 0 study.
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable.
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured.
* Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression for ≥ 1 month after treatment of the brain metastases.
* Patients with a prior or concurrent malignancy are eligible for this trial if, in the judgement of the principal investigator, the malignancy and its treatment do not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better.
* The effects of pidnarulex on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) 14 days prior to study entry and for the duration of study participation and for at least 6 months after the last dose of study drug. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Women should not breastfeed while taking pidnarulex and for 6 months after cessation of treatment. Men treated or enrolled on this protocol must also agree to use adequate contraception 14 days prior to the study, for the duration of study participation, and 6 months after completion of pidnarulex administration.
* Willingness to provide blood and biopsy samples for research purposes.
* Ability to understand and the willingness to sign a written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants.

Exclusion Criteria:

* Patients must have recovered from clinically-significant adverse-events of their most recent cancer immunotherapy to grade 1 or less (with the exception for alopecia or lymphopenia).
* Eligibility of subjects receiving any medications or substances known to affect or with the potential to affect the activity of pidnarulex will be determined based on their potential to interact with the CYP3A4 isozyme. Specifically, subjects taking strong CYP3A4 inhibitors or strong CYP3A4 inducers will be excluded from participation in the trial. A list of agents that interact with CYP450 isoenzymes is provided. For medications or substances not listed, or in cases of uncertainty, the principal investigator may consult with a medical expert or a pharmacologist to make an informed decision regarding eligibility.
* History of allergic reactions attributed to inactive ingredients in the drug product.
* Patients with uncontrolled intercurrent illness or any other significant condition(s) that would make this protocol unreasonably hazardous.
* Pregnant and lactating women are excluded from this trial. The exclusion is based on the potential risk of adverse effects of pidnarulex on fetal development and newborn health. The safety of pidnarulex has not been established in pregnant or lactating women, and there is a possibility that the drug could cause harm to the developing fetus or be transferred to the infant through breast milk. Additionally, the physiological changes that occur during pregnancy and lactation could alter the pharmacokinetics and pharmacodynamics of pidnarulex, leading to unpredictable drug exposure and efficacy.
* Patients with chronic, active HBV or HCV infections that require ongoing antiviral treatment will be excluded from the trial. This exclusion is due to the potential for drug interactions with the study medication and the risk of exacerbating liver disease.
* Patients with cirrhosis, regardless of the etiology, will be excluded from participation in the trial. This is due to the increased risk of complications and adverse events associated with the study medication in this population.
* Presence of known photosensitivity disorders (xeroderma pigmentosa, porphyria etc.). Patients who do not agree to use sunglasses and sun blocker (with sun protection factor 50 [SPF50] to ultraviolet B [UVB] and a high degree of protection against ultraviolet A [UVA]) if exposed to sunlight during the course of the study and for 3 months after the last dose are not eligible. Appropriate sunscreen products will be provided. Patients who plan to use sun beds or tanning booths during the course of the study and within 3 months after the last dose are not eligible.
* Active ocular surface disease at baseline (based on ophthalmological evaluation).
* History of cicatricial conjunctivitis (as evaluated by an ophthalmologist).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
RAD51 response | Up to 3 years
  Will be defined as at least 5 percent of cells with at least 5 positive foci per nucleus. Will target a 30% Rad51 response rate. Will be compared descriptively across the 2 cohorts, with and without homologous repair deficiency mutations.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 3 years
  Will be summarized using Common Terminology Criteria for Adverse Events version 5.0.
Overall response | From the time measurement criteria are met for complete response or partial response until the first date that recurrent or progressive disease is objectively documented; assessed up to 3 years
Pharmacokinetics (PK) | At baseline, post-infusion on cycle (C) 1 day (D) 1, before the biopsy on C1D2, pre-infusion and post-infusion C1D8, and C1D15
  PK will be measured using plasma.
Deoxyribonucleic acid (DNA) damage and repair signaling markers | Up to 3 years

OTHER OUTCOMES:
Genomic alterations | Up to 3 years
  Will be measured using circulating tumor DNA. Will be assessed using non-parametric analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Jibran Ahmed, Principal Investigator — National Cancer Institute LAO
Locations (1):
- National Cancer Institute Developmental Therapeutics Clinic, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm